CLINICAL TRIAL: NCT05032222
Title: The Role of "Hypospadias Objective Scoring Evaluation" (HOSE) and Uroflowmetry in Evaluation of Successful Hypospadias Repair
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Mohammad Alaa Ezzat (Other)
Responsible Party: Sponsor-Investigator, Mohammad Alaa Ezzat, Resident, Assiut University
Organization: Assiut University (Other)
Other Study IDs: Hypospadias repair evaluation
Record Dates: First submitted 2021-08-27; First posted 2021-09-02 (Actual); Last update posted 2021-09-27 (Actual); Status verified 2021-09

CONDITIONS: Hypospadias
MeSH Terms: conditions — Hypospadias

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Uroflowmetry — Diagnostic test

SUMMARY:
Hypospadias is a common anomaly of the male genitalia affecting 0.4-8.2 of 1000 live male babies and varies considerably in severity. The position of the urethral meatus can be classified as anterior or distal (glandular, coronal, or subcoronal; 60-65% of cases), middle (midpenile; 20-30% of cases), or posterior or proximal (posterior penile, penoscrotal, scrotal, or perineal; 10-15% of cases). The subcoronal position is the most common. Most cases are mild and surgical correction is undertaken mostly for cosmetic reasons at the request of the parents or on advice of the pediatrician or surgeon.

Functional success of hypospadias repair depends on the creation of a uniform and adequate caliber urethra up to the meatus. Accordingly, meatal stenosis and urethral stricture are the important complications of surgery, others include urethrocutaneous fistula, diverticula, skin flap necrosis and persistent chordee. Although functional assessment of the repair is possible by observation of the urinary stream and voiding cystourethrography, uroflowmetry is considered to be a more objective tool, especially for the detection of a subclinical urethral stricture. Reports of the results of hypospadias surgery commonly focus on the cosmetic results and incidence of obvious complications, as urethrocutaneous fistulas, and symptomatic urethral Strictures. Few have emphasized the role of uroflowmetry in the postoperative evaluation of children with hypospadias to detect asymptomatic strictures and, despite the simplicity and non-invasive nature of this test, it has not become standard or widely accepted.

We evaluate AUUH experience by use of 'hypospadias objective scoring evaluation' HOSE and uroflowmetry after hypospadias repair. The HOSE is a validated scoring system that incorporates the evaluation of meatal location and shape, urinary stream, straightness of erection, presence and complexity of urethral fistula. The minimum total score is 5, and the maximum total score is 16. The point score is graded as either acceptable or not.

ELIGIBILITY:
Inclusion Criteria:

1. More than six months after last hypospadias repair.
2. Toilet trained children.
3. Patients less than 18 years old.
4. Successful repair of hypospadias with HOSE score more than 10 decided by one of the experts in pediatric urology.

Exclusion Criteria:

1. Patient not welling to participate in our study.
2. Within six months of last hypospadias repair.
3. Patient had urethral intervention within 3 months.
4. Children with any associated neurological or urological abnormality related to the bladder, which could potentially affect flow pattern.

Ages: 6 Months to 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes
Study Population: All cases that fulfil the selection criteria that will be followed up in the department of Assiut university hospital (non probability sample size) with Confidence Level 90 % , Population Size 10000 , Margin of Error 8 % with expected size of 105 patients starting from 01/04/2021 to 1/04/2022.
Sampling Method: Non-Probability Sample
Enrollment: 105 (Estimated)
Dates: Start 2021-05-01 (Actual); Primary Completion 2023-05-01 (Estimated); Study Completion 2023-05-01 (Estimated)

PRIMARY OUTCOMES:
Number of patients show Change of the maximum flow rate, average flow rate (Qav), total voided volume, PMR and voiding time from normal values. | Within 5 years post operative
  Number of patients show Change of the maximum flow rate, average flow rate (Qav), total voided volume, PMR and voiding time from normal values.
Number of patients in each Type of the curve of the uroflowmetry. | Within 5 years postoperative
  Number of patients in each Type of the curve of the uroflowmetry.
Finding correlation between the results of uroflowmetry and HOSE score. | Within 5 years postoperative
  Finding correlation between the results of uroflowmetry and HOSE score.

CONTACTS AND LOCATIONS:
Overall Officials: Hisham M Hammoda, Professor, Study Director — Assiut University; Amr H Abo fadan, Lecturer, Study Director — Assiut University; Mahmoud F Ali, Lecturer, Study Director — Assiut University
Locations (1):
- Assiut university hospital, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Olsen LH, Grothe I, Rawashdeh YF, Jorgensen TM. Urinary flow patterns in infants with distal hypospadias. J Pediatr Urol. 2011 Aug;7(4):428-32. doi: 10.1016/j.jpurol.2010.05.013. Epub 2010 Jul 2. PMID 20598640
- [Background] Page RE, Akin Y. Assessment of urine flow in hypospadias. Br J Plast Surg. 1978 Oct;31(4):313-6. doi: 10.1016/s0007-1226(78)90117-0. No abstract available. PMID 152135
- [Background] Toguri AG, Uchida T, Bee DE. Pediatric uroflow rate nomograms. J Urol. 1982 Apr;127(4):727-31. doi: 10.1016/s0022-5347(17)54018-5. No abstract available. PMID 7069841
- [Background] Gonzalez R, Ludwikowski BM. Importance of urinary flow studies after hypospadias repair: a systematic review. Int J Urol. 2011 Nov;18(11):757-61. doi: 10.1111/j.1442-2042.2011.02839.x. Epub 2011 Aug 30. PMID 21883491
- [Background] Kaya C, Kucuk E, Ilktac A, Ozturk M, Karaman MI. Value of urinary flow patterns in the follow-up of children who underwent Snodgrass operation. Urol Int. 2007;78(3):245-8. doi: 10.1159/000099346. PMID 17406135
- [Background] Holmdahl G, Karstrom L, Abrahamsson K, Doroszkiewicz M, Sillen U. Hypospadias repair with tubularized incised plate. Is uroflowmetry necessary postoperatively? J Pediatr Urol. 2006 Aug;2(4):304-7. doi: 10.1016/j.jpurol.2005.11.018. Epub 2006 Mar 30. PMID 18947626
- [Background] Garignon C, Chamond C, Lefebure B, Halim Y, Mitrofanoff P, Liard A. [Uroflowmetric functional evaluation of modified Duplay procedure in hypospadias surgery]. Prog Urol. 2004 Dec;14(6):1199-202; discussion 1202. French. PMID 15751419
- [Background] Jayanthi VR, McLorie GA, Khoury AE, Churchill BM. Functional characteristics of the reconstructed neourethra after island flap urethroplasty. J Urol. 1995 May;153(5):1657-9. PMID 7715002
- [Background] Scarpa MG, Castagnetti M, Berrettini A, Rigamonti W, Musi L. Urinary function after Snodgrass repair of distal hypospadias: comparison with the Mathieu repair. Pediatr Surg Int. 2010 May;26(5):519-22. doi: 10.1007/s00383-010-2569-6. Epub 2010 Feb 19. PMID 20169443
- [Background] Wolffenbuttel KP, Wondergem N, Hoefnagels JJ, Dieleman GC, Pel JJ, Passchier BT, de Jong BW, van Dijk W, Kok DJ. Abnormal urine flow in boys with distal hypospadias before and after correction. J Urol. 2006 Oct;176(4 Pt 2):1733-6; discussion 1736-7. doi: 10.1016/S0022-5347(06)00614-8. PMID 16945635
- [Background] Tuygun C, Bakirtas H, Gucuk A, Cakici H, Imamoglu A. Uroflow findings in older boys with tubularized incised-plate urethroplasty. Urol Int. 2009;82(1):71-6. doi: 10.1159/000176029. Epub 2009 Jan 20. PMID 19172101
- [Background] Eassa W, Brzezinski A, Capolicchio JP, Jednak R, El-Sherbiny M. How do asymptomatic toilet-trained children void following tubularized incised-plate hypospadias repair? Can Urol Assoc J. 2012 Aug;6(4):238-42. doi: 10.5489/cuaj.12029. PMID 23093529